CLINICAL TRIAL: NCT01662362
Title: Abbott ESA Chagas Assay Post-Market Study
Acronym: ESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diagnostics Division (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 7B5-02-10P02-01
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-01

CONDITIONS: Chagas Disease
Keywords: Chagas Disease; Trypanosoma cruzi; American trypanosomiasis; South American trypanosomiasis; kissing bugs; reduviid bugs
MeSH Terms: conditions — Chagas Disease | interventions — Biological Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testing Donor Specimens with ESA Chagas (Other): Test blood donor specimens that are ABBOTT PRISM Chagas Repeatedly Reactive with ESA Chagas. Donors will be asked to return for a follow-up blood draw.
  Interventions: Device: Testing Donor Specimens with ESA Chagas

INTERVENTIONS:
Device: Testing Donor Specimens with ESA Chagas — Donors will be asked to return for a follow-up blood draw.
  Other Names: ABBOTT ESA Chagas (ESA Chagas) assay; List Number: 8L34

SUMMARY:
The study is conducted to meet an FDA post market commitment to collect and report data on the performance of the ESA Chagas assay. A minimum of 50 donor specimens that are FDA-licensed ABBOTT PRISM Chagas repeatedly reactive (RR)will be tested with the ABBOTT ESA Chagas assay. In addition, minimum of 300 ABBOTT PRISM Chagas nonreactive (NR) unidentified donor specimens will be tested with ABBOTT ESA Chagas assay.

DETAILED DESCRIPTION:
ABBOTT ESA Chagas testing will be performed at a minimum of two blood donor centers. Testing will be performed using the FDA-licensed ESA Chagas assay and will be performed in accordance with the ESA Chagas package insert. ABBOTT PRISM Chagas repeatedly reactive blood donor specimens identified by U.S. blood donor centers, as part of the routine blood donation process, will be tested with the FDA-licensed ESA Chagas. Specimens will also be tested with radioimmune precipitation assay (RIPA) for antibody to T. cruzi, a laboratory developed test, and the FDA-licensed ORTHO T. cruzi ELISA. The donor centers will contact the donors and request the donor to return to complete a questionnaire and provide a follow-up specimen.

In addition, a minimum of 300 blood donor specimens with ABBOTT PRISM Chagas nonreactive results will also be tested with ESA Chagas. These specimens will be unidentified, leftover specimens from routine donor testing and not individually identifiable. Specimens that are positive or indeterminate with ESA Chagas will be further tested with RIPA.

ELIGIBILITY:
PRISM Chagas Repeatedly Reactive Donor Specimens

Inclusion Criteria:

* Blood donor specimen documented as PRISM Chagas repeatedly reactive

Exclusion Criteria:

* None

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stramer, Ph.D., Principal Investigator — American National Red Cross; Sharon Gordon, MS, MBA, MT, Principal Investigator — LifeSource
Locations (2):
- United States (2):
  - LifeSource, Rosemont, Illinois
  - American Red Cross, Gaithersburg, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Testing Donor Specimens With ESA Chagas
Started | 63
Completed | 25
Not Completed | 38
Not completed — Lost to Follow-up | 38

BASELINE CHARACTERISTICS:
Population: Donor specimens PRISM Chagas Repeatly Reactive
Arm/Group | Testing Donor Specimens With ESA Chagas
Number analyzed (Participants) | 63
Age, Customized [Number; unit: participants] — Routine whole blood donors
  participants
    >= 18 years | 19
    Unknown | 44
Sex/Gender, Customized [Number; unit: participants]
  Male | 9
  Female | 10
  Unknown | 44
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: ESA Chagas Testing of US Blood Donor Specimens Repeatedly Reactive by ABBOTT PRISM Chagas
Time Frame: Up to six months
Measure: Number (95% Confidence Interval); unit: percent agreement to RIPA
Arm/Group | Testing Donor Specimens With ESA Chagas
Number analyzed (Participants) | 63
percent agreement to RIPA | 92.06 [82.44 to 97.37]

2. Secondary Outcome: ESA Testing of Preselected Donor Specimens Nonreactive by ABBOTT PRISM Chagas
Time Frame: Up to six months
Measure: Number (95% Confidence Interval); unit: percentage of specimens ESA negative
Groups:
- Testing Donor Specimens With ESA Chagas: Test blood donor specimens that are ABBOTT PRISM Chagas Nonreactive with ESA Chagas. These specimens will be unidentified specimens from routine donor testing and not individually identifiable. Specimens that are positive or indeterminate with ESA Chagas will be further tested with RIPA.
Arm/Group | Testing Donor Specimens With ESA Chagas
Number analyzed (Participants) | 300
percentage of specimens ESA negative | 99.00 [97.11 to 99.79]

ADVERSE EVENTS:
Arm/Group | Testing Donor Specimens With ESA Chagas
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days